CLINICAL TRIAL: NCT03093597
Title: Evaluating Skin Barrier Biophysical Properties and Clinical Appearance After Moisturizer Use in Patients With Dry Skin
Brief Title: Skin Barrier Biophysical Properties and Clinical Appearance After Moisturizer in Dry Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1701110479
Record Dates: First submitted 2017-03-23; First posted 2017-03-28 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2017-01

CONDITIONS: Xerosis; Xerosis Cutis; Dry Skin; Eczema
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- virgin coconut oil (Active Comparator): All subjects will apply virgin coconut oil to a previously randomize section of the skin on the left or right forearm.
  Interventions: Other: virgin coconut oil
- virgin jojoba oil (Active Comparator): All subjects will apply virgin jojoba oil to a previously randomize section of the skin on the left or right forearm
  Interventions: Other: virgin jojoba oil
- virgin almond oil (Active Comparator): All subjects will apply virgin almond oil to a previously randomize section of the skin on the left or right forearm
  Interventions: Other: virgin almond oil
- white petrolatum ointment (Active Comparator): All subjects will apply white petrolatum ointment to a previously randomize section of the skin on the left or right forearm.
  Interventions: Other: white petrolatum ointment

INTERVENTIONS:
Other: virgin coconut oil — One of the four locations (right proximal forearm, right distal forearm, left proximal forearm, left distal forearm) on the forearm will be selected to receive virgin coconut oil application twice daily for 2 weeks.
  Arms: virgin coconut oil
Other: virgin jojoba oil — One of the four locations (right proximal forearm, right distal forearm, left proximal forearm, left distal forearm) on the forearm will be selected to receive virgin jojoba oil application twice daily for 2 weeks.
  Arms: virgin jojoba oil
Other: virgin almond oil — One of the four locations (right proximal forearm, right distal forearm, left proximal forearm, left distal forearm) on the forearm will be selected to receive virgin almond oil application twice daily for 2 weeks.
  Arms: virgin almond oil
Other: white petrolatum ointment — One of the four locations (right proximal forearm, right distal forearm, left proximal forearm, left distal forearm) on the forearm will be selected to receive white petrolatum ointment application twice daily for 2 weeks.
  Arms: white petrolatum ointment

SUMMARY:
The purpose of the study is to compare the changes in the appearance of dry skin after the use various moisturizers: white petrolatum ointment, coconut oil, jojoba oil, and almond oil in patients with dry skin.

DETAILED DESCRIPTION:
The goal of this study is to compare how the appearance of dry skin changes before and after the use of following moisturizers: white petrolatum, coconut oil, jojoba oil and almond oil). Up to 40 subjects from Banner-University Medical Center/University of Arizona dermatology clinics and University of California, Davis dermatology clinics (up to 20 subjects per site) who have dry skin will be enrolled in this study and randomized to receive the four moisturizers on four locations on their forearms.There will be a total of 3 study sessions: baseline, and approximately 1 and 2 weeks for follow up assessment. At each visit, dry skin severity will be evaluated by a trained observer using a validated Dry Skin Score, skin barrier biophysical properties (transepidermal water loss and hydration) will be measured, and digital photos of the test sites will be taken for image analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, at least 18 years of age
2. Subject must receive a diagnosis of dry skin by a dermatologist.
3. Subject must be able to comprehend and read the English language.

Exclusion Criteria:

1. Subjects who do not fit the inclusion criteria.
2. Subjects unable to or unwilling to comply with the study procedures
3. Prior known allergy to white petrolatum, coconut oil, almond oil, or jojoba oil.
4. People who have used products containing white petrolatum, jojoba oil, coconut oil, or almond oil within the past week.
5. People with a known diagnosis of ichthyosis.
6. A subject who, in the opinion of the investigator, will be un-cooperative or unable to comply with study procedures.
7. Subject unable to speak or read the English language, since all consents and instructions will be provided in English.
8. Those that are prisoners or cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
The appearance of xerosis | 14 days
  The clinical severity of xerosis of the 4 location will be graded by a trained observed using a previously validated Dry Skin Scale and by analysis of the digital photos.

OTHER OUTCOMES:
Skin barrier biophysical properties of xerosis | 14 days
  Transepidermal water loss (TEWL) and stratum corneum hydration status will be measured using hand-held, noninvasive, skin barrier measuring devices (Tewameter and moistureMeter)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Y Shi, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona, Banner-University Medical Center, Tucson, Arizona
  - University of California, Davis, Sacramento, California

IPD SHARING:
Plan to Share IPD: No